CLINICAL TRIAL: NCT05937048
Title: Coagulation Parameters With Albumin in Decompensated Cirrhosis (CoPA-D): An Open-label Randomized Control Trial
Brief Title: Coagulation Parameters With Albumin in Decompensated Cirrhosis (CoPA-D).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-55
Record Dates: First submitted 2023-02-20; First posted 2023-07-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-06

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — Albumins; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin (Experimental): 20% human albumin solution infusion, to raise and maintain serum albumin levels above 3.0 g/dl. Human albumin solution will be given to those enrolled in the study having serum albumin levels ≤ 3 g/dl to maintain the serum albumin levels above 3 g/dl.
  Interventions: Biological: Albumin
- Standard of Care (Active Comparator): Standard treatment that the patient would receive had they not been included in the trial.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: Albumin — 20% human albumin solution infusion, to raise and maintain serum albumin levels above 3.0 g/dl. Human albumin solution will be given to those enrolled in the study having serum albumin levels ≤ 3 g/dl to maintain the serum albumin levels above 3 g/dl.
  Arms: Albumin
Other: Standard of Care — Standard treatment that the patient would receive had they not been included in the trial.
  Arms: Standard of Care

SUMMARY:
Albumin is commonly used plasma expander in patients of decompensated cirrhosis and has been found to have many beneficial effects, with few studies showing that maintenance of serum albumin levels above 3 g/dl has improved outcomes and mortality leading to widespread utilization in patients with cirrhosis of the liver.

While 20% human albumin solution has been subject to in-depth analysis along several fronts, it's effects on coagulation parameters is unknown. With cirrhosis being a state of dysregulated clotting and bleeding, it is imperative to know the effects of such a widely used plasma expander on coagulation.

The aim of this study is to evaluate the effects of albumin on coagulation parameters in patients of decompensated cirrhosis.

DETAILED DESCRIPTION:
Aim and Objective:

To study the effects of 20% human albumin infusions on coagulation parameters in patients with decompensated cirrhosis of the liver.

Methodology:

- Study population: All patients aged ≥ 18 years and ≤ 70 years admitted in Institute of Liver and Biliary Sciences, New Delhi with decompensated cirrhosis of any cause and S. Albumin ≤ 2.5 g/dl upon presentation and are giving written consent for participation in the study.

* Study design - Single center, Open label, Randomized controlled trial
* Study period - 1 year
* Monitoring and assessment -
* ABG prior to enrollment
* Investigations - tests performed on Day 0, 1, 3, 5 and 7 or till discharge (whichever is earlier)

  * Routine: CBC, RFT, LFT, apTT, PT/INR, CXR
  * Coagulation parameter: ROTEM (EXTEM, FIBTEM), Fibrinogen
  * Inflammatory markers: ESR, CRP, IL-6, TNF-⍺
  * Endothelial dysfunction: vWF, ADAMTS-13
  * Cardiac function: NT-proBNP, PRA
  * 2 D Echo,PFT with DLCO will be done at 0,1 and 7 days.
* Statistical Analysis:

The data will be represented as mean±SD. The categorical data will be analysed using Chi-square test. The continuous data will be analysed by student T test, or Mann-Whitney test, whichever is applicable. Besides this, Cox regression will be applied to analyse the variables. For all tests, p≤ 0.05 will be considered statistically significant.

* Adverse effects
* Allergic reactions to albumin.
* Features of symptomatic volume overload.
* Stopping rule
* Day 7, or discharge (whichever is earlier)
* Allergic reaction to albumin
* Features of symptomatic volume overload
* Variceal bleeding
* Requirement of coagulation correct

Expected outcome of the project:

Derangement of ROTEM in the group of patients receiving human albumin solution

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 70 years
* Decompensated cirrhosis of any cause
* S. Albumin ≤ 2.5 g/dl upon presentation
* Written informed consent

Exclusion Criteria:

* Patients of ACLF
* Patients admitted with proven indications for albumin (SBP, HRS, LVP)
* Advanced HCC
* Presence of hypotension
* PF ratios ≤ 300 mmHg on arterial blood gas
* IVC Collapsibility Index < 20%
* Albumin infusion within the past 3 weeks
* Post liver transplant patients
* AKI or CKD
* Known or suspected cardiac dysfunction
* Acute GI Bleed
* Severe Anemia
* Pregnant women
* PLHA
* Severe psychiatric disorders
* Lack of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Change in ROTEM based coagulation parameters with albumin infusion in decompensated cirrhotic patients. | 3 days
  ROTEM based parameters includes CT,CFT,A10,A20,MCF (EXTEM). CT,CFT,A10,A20 (FIBTEM)

SECONDARY OUTCOMES:
Changes in inflammatory parameters like ESR. | 3 days
Changes in inflammatory parameters like CRP. | 3 days
Changes in inflammatory parameters like IL-6 | 3 days
Changes in inflammatory parameters like TNF-alpha. | 3 days
Changes in endothelial dysfunction like VWF. | 3 days
Changes in endothelial dysfunction like ADAMTS-13. | 3 days
Effect on pulmonary function by Pulmonary function test | 3 days
Effect on renal function by s.creatinine. | 3 days
Adverse effects of Human Albumin Solution | 3 days
Change in the albuminome in both the groups | 3 days
  Albumin bound metabolites and lipids will be studied and the effect of albumin infusion on this albuminome.
Duration of hospital stay | 28 days
Mortality at 28 days | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided